CLINICAL TRIAL: NCT05569928
Title: In Vivo Metabolism of apoB-containing Lipoproteins in ANGPTL3 Deficient Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marcello Arca (Other)
Collaborators: Pfizer (Industry); Göteborg University (Other); University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Marcello Arca, Full Professor, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0061/2022
Record Dates: First submitted 2022-09-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Familial Hypobetalipoproteinemia; Familial Hypobetalipoproteinemia - Heterozygous Form
Keywords: FHBL2; ANGPTL3; Kinetic study; ApoB lipoprotein metabolism
MeSH Terms: conditions — Hypobetalipoproteinemias; Hypobetalipoproteinemia, Familial, 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Homozygous FHBL2 subjects (Active Comparator)
  Interventions: Other: Administration of deuterated compounds for kinetic study
- Heterozygous FHBL2 carriers (Active Comparator)
  Interventions: Other: Administration of deuterated compounds for kinetic study
- ANGPTL3 wild-type Campodimele residents (Active Comparator)
  Interventions: Other: Administration of deuterated compounds for kinetic study

INTERVENTIONS:
Other: Administration of deuterated compounds for kinetic study — Participants will be submitted to a standardized oral-fat load and kinetic study will be performed

SUMMARY:
Rationale. ANGPTL3 has been identified as important regulator of lipolysis as well as a determinant of plasma levels of apolipoprotein B-containing lipoproteins. However, the precise mechanisms by which ANGPTL3 influences the flux of apoB particles transiting from the VLDL into LDL density range or affect LDL synthesis by modulating chylomicron remnants removal are unclear. It has been reported that the genetically determined ANGPTL3 absence or deficit is linked to lower plasma levels of apoB-containing lipoproteins. Therefore, a way to address the action of ANGPTL3 is to evaluate the in vivo lipoprotein metabolism in subjects carrying genetic mutations lowering ANGPTL3 as compared to normal controls.

Overall goal. The aim of this proposal is to uncover the role of ANGPTL3 in chylomicron, VLDL and LDL metabolism in humans (with a particular focus on its impact on the VLDL to LDL conversion pathway) using well-established in vivo lipoprotein kinetic methodologies.

Target population. For the present study, we will recruit subjects carrying the loss-of function mutation S17X in ANGPTL3 gene. Of them, 4 will be homozygotes, showing undetectable plasma levels of ANGPTL3 and hypobetalipoproteinemia and 8 will be heterozygotes with low ANGPTL3 plasma levels (<150 ng/ml), low TG (<120mg/dl) and LDL-C <160 mg/dl. Gender, age and BMI matched controls (n= 8) with plasma TG<180 mg/dl and LDL-C <160 mg/dl, and no known factors perturbing lipid metabolism will also be recruited. Cases and controls will be recruited from the Campodimele population.

Methods. Subjects will receive a 500 mg injection of deuterated glycerol to assess triglyceride kinetics, and an injection of deuterated leucine (7 mg/kg body weight) to assess the kinetics of apoB100, apoB48, apoC-III, and apoE. To evaluate chylomicron metabolism, subjects will be served a standard fat rich meal that contain 927 kcal (59.5 % fat, 24.4 % carbohydrate and 15.5 % protein) 2 hrs after injection of isotopes. Blood samples will be taken at frequent time points for 8 hrs followed by further blood samples collected next morning (24 hours) and on days 2, 3 and 4 after tracer administration. Chylomicrons, VLDL1, VLDL2, IDL and LDL will be isolated in a well-established stepwise centrifugal procedure. The concentrations of lipids and apolipoproteins will be determined using immunoassay and mass spectrometry in whole plasma and in lipoprotein fractions at each time point in the metabolic protocol. Isotope enrichment in apoproteins and lipids (triglycerides) will be performed using GC/MS.

Assessment. The main kinetic parameters derived from multicompartmental models will be:

1. Production and fractional clearance rates for apoB48-containing particles in chylomicrons, VLDL1, VLDL2, and for apoB100-containing particles in VLDL1, VLDL2, IDL and LDL.
2. Lipolysis rates for TG in VLDL1 and VLDL2.
3. Rates of conversion of chylomicrons to VLDL1 and VLDL2, rates of conversion of VLDL1 to VLDL2 to IDL and to LDL.

DETAILED DESCRIPTION:
Working hypothesis

The overall working hypothesis is that the normal physiological action of ANGPTL3 is to slow lipolysis and inhibit remnant clearance by the liver. In this way, the protein causes an increase in the flux of apoB particles transiting from the VLDL into LDL density range, resulting in a net increase in LDL production. In previous studies we observed that the extent of conversion of VLDL to IDL and then LDL varies from 25% to 75%.2 Where and how ANGPTL3 might act remains to be discovered. A comparison of the rates of VLDL1 and VLDL2 production, rates of lipolysis of these particles, and the amount of apoB converted to IDL and then LDL in control subjects and those heterozygous and homozygous for ANGPTL3 loss-of-function (LOF) variants will enable us to delineate where ANGPTL3 acts, and possibly reveal a gene-dose related effect.

Alternative hypotheses will also be explored including the possibility that accelerated chylomicron lipolysis in ANGPTL3 LOF carriers leads to a subnormal amount of dietary triglyceride being delivered to the liver which as a result impairs VLDL assembly and secretion. This would imply that the hypobetalipoproteinaemia phenotype is primarily due to an abnormality in hepatic production. Or, as recently suggested from studies in familial hypercholesterolemia, that there is a stimulation of LDL catabolism when ANGPTL3 activity is reduced.

Primary Objectives

The primary objectives are to investigate in subjects heterozygous and homozygous for ANGPTL3 LOF variants compared to matched controls the:

* Kinetics of apoB48 in chylomicrons and their remnants in light of our earlier investigations that revealed dramatic reductions in post-prandial chylomicronaemia in homozygous LOF carriers.4
* Kinetics of apoB100 in VLDL1, VLDL2, IDL and LDL. This will reveal the basis for the hypobetalipoproteinaemia seen in this condition 4-6 and clarify how partial or complete loss of ANGPTL3 leads to lower levels of VLDL, remnants, and LDL.
* Kinetics of TG in VLDL1 and VLDL2. This will reveal how lipolysis is altered when ANGPTL3 action is impaired or absent.

Secondary Objectives

Our secondary objectives are to investigate:

* The impact of ANGPTL3 on the kinetics of the key regulatory apolipoproteins apoC-III and apoE, since apoC-III has been reported to be lower in concentration when ANGPTL3 is reduced.
* The detailed composition of apoB-containing lipoprotein species. We will explore the proteomic and lipidomic profiles of chylomicrons, VLDL1, VLDL2, IDL and LDL in this unique cohort to understand further the compositional signatures in this specific 'low ASCVD risk' condition.

Experimental Design and Approach Subjects recruitment: Subjects will be recruited on the basis of their known status for the S17X LOF variant. The individuals are inhabitants of the Campodimele village, near Rome, Italy. The investigators have over many years established a close and mutually valued connection with the people of Camapodimele and have published key characteristics of the lipid phenotype that is exhibited by those carrying the ANGPTL3 LOF, which is a profound combined hypolipidemia associated with reduced plasma levels of total cholesterol, TG, VLDL-TG and cholesterol, LDL cholesterol, apoB, and a blunted post-prandial triglyceride response to a test fat meal. Our plan is to recruit the 4 available homozygotes and identify 6-8 heterozygotes who exhibit low ANGPTL3 plasma levels (<150ng/ml) and low TG (<120mg/dl). Age and sex matched healthy controls (n=6-8) with no known factors perturbing lipid metabolism will also be recruited from the Campodimele population.

Metabolic protocol: The investigators have developed and validated novel methods allowing to simultaneously follow the kinetics of TGs in large VLDL1 and smaller VLDL2, apoB48 in chylomicrons, VLDL1 and VLDL2, apoB100 in VLDL1, VLDL2, IDL and LDL, and the production and catabolic rates for apoC-III and apoE. Subjects will receive a 500 mg injection of deuterated glycerol to assess triglyceride kinetics, and an injection of deuterated leucine (7 mg/kg body weight) to assess the kinetics of apoB100, apoB48, apoC-III, and apoE. To evaluate chylomicron metabolism, subjects will be served a standard fat rich meal that contain 927 kcal (59.5 % fat (68 g), 24.4 % carbohydrate (63 g) and 15.5 % protein (40 g) 2 hrs after injection of isotopes. Blood samples will be taken at frequent time points for 8 hrs followed by further blood samples collected next morning (24 hours) and on days 2, 3 and 4 after tracer administration. The total blood volume to be withdrawn over the period of the kinetic study (about 350 ml) has been reduced in recognition that some of the subjects (homozygotes in particular) are elderly. (This volume of blood donation is considered acceptable and is below what has been collected in earlier clinical studies in this population). The reduction in blood drawn does not alter our ability to derive the full set of kinetic parameters - The investigators will make best use of the highly sensitive analytical techniques. Dr Arca's clinical team will perform the metabolic protocol on site at special clinical premises in Campodimele. Samples will be taken to his laboratory in Rome for aliquoting and shipment. Lipoprotein isolation: Isolation of lipoprotein fractions for kinetic analysis is time consuming and requires specialised equipment (ultracentrifuges) and considerable expertise; isolating TRL fractions from subjects with low plasma TG is even more challenging. Preparation of lipoprotein fractions will therefore be undertaken in the laboratory of Dr Taskinen in Helsinki (after shipment on ice from Rome). Chylomicrons, VLDL1, VLDL2, IDL and LDL will be isolated in a well-established stepwise centrifugal procedure. First, total TRL will be concentrated by ultracentrifugation (d <1.006 g/ml for 18 hrs) and then this 'top' fraction will be harvested and used to isolate chylomicrons (Sf >400), VLDL1 (Sf 60-400), and VLDL2 (Sf 20-60) by density gradient ultracentrifugation. The d>1.006 g/ml ('bottom') fraction will be used to separate IDL and LDL in further sequential centrifugation steps. These methods are employed routinely in the Helsinki lab. The isolated lipoprotein fractions are then prepared for transfer to Gothenburg for enrichment analyses. This preparation involves measurements of TG, cholesterol, phospholipids and protein concentration, and delipidation, precipitation and measurement of apoB. Analyses of enrichments of isotopes in apoproteins and lipids, and mathematical modelling: The next step in the kinetic investigation is the analysis of the enrichment of stable isotopes using highly sensitive mass spectrometry methods. The concentrations of lipids and apolipoproteins (apoB100, apoB48, apoC-III and apoE) will be determined using immunoassay and mass spectrometry techniques in whole plasma and in lipoprotein fractions at each time point in the metabolic protocol. Isotope enrichment in apoproteins and lipids (triglycerides) will be performed using GC/MS. All of these methods, including sample transfers, are robust and well established in the Helsinki and Gothenburg labs, and have been the subject of a series of publications. The isotope enrichment results and TG/apoprotein concentrations in all the isolated fractions form the data set on which the multicompartmental modelling is conducted. The investigators have successfully developed and applied our models to data derived from subjects with a variety of conditions (hypertriglyceridemia, hypotriglyceridaemia, diabetes) as well as on and off lipid-lowering treatment. The models are applicable to all settings encountered and have generated novel insights into lipoprotein metabolism.12x-14 Kinetic parameters derived from multicompartmental models are: Production rates for apoB48 particles in the chylomicron, VLDL1 and VLDL2 fractions. Production rates for apoB100 in VLDL1, VLDL2, IDL and LDL. Lipolysis rates for TG in VLDL1 and VLDL2 Fractional clearance rates for apoB48-containing particles in chylomicrons, VLDL1, VLDL2, and for apoB100-containing particles in VLDL1, VLDL2, IDL and LDL. Rates of conversion of chylomicrons to VLDL1 and VLDL2, rates of conversion of VLDL1 to VLDL2 to IDL and to LDL. Production and clearance rates of apoC-III and apoE.

Main Outcome Measures and Study Deliverables. How ANGPTL3 regulates lipoprotein metabolism in humans is unknown and, therefore, it is important to keep an open mind as to its precise mode of action on apoB and TG kinetics as explored in this study. Our working hypothesis based on observations to date in LOF carriers is that it has an impact on all apoB-containing lipoproteins that is distinct from other regulatory factors such as those that alter lipoprotein production - microsomal triglyceride transfer (MTP) protein activity or mutations that inhibit VLDL1 assembly (TM6SF2), or those that alter lipoprotein receptor-mediated clearance such as PCSK9.

The investigators have recently published research of factors that alter apoB and TG production such as TM6SF2, PNPLA3 and the role of PCSK9 in controlling the catabolism of apoB-containing lipoproteins. Further, and importantly, the investigators are just completing a kinetic study in a group of apoCIII LOF carriers who exhibit low TG levels and other phenotypic traits comparable to those seen in ANGPTL3 LOF (as yet unpublished). The availability of these comparator studies provides a metabolic background against which we can evaluate the specific actions of ANGPTL3.

The primary evaluation will focus on the differences in VLDL1, VLDL2, IDL and LDL clearance rates, the rates of TG lipolysis in VLDL1 and VLDL2, and the rates of conversion of VLDL1/ VLDL2 to IDL and LDL in the homozygous S17X carriers compared to heterozygotes and controls. The key research question is "does ANGPTL3 deficiency or absence result in increased lipolysis and increased fractional clearance rates for VLDL2 and IDL (the precursors of LDL) which then leads to reduced intravascular generation of LDL particles, and possibly reduction in the circulating level of remnant lipoproteins". the investigator will also explore a potential gene-dose effect by including heterozygotes in the statistical analysis. The key kinetic parameters will be tested in ANOVA models, with inclusion of potential confounding factors such as sex and BMI.

the secondary hypothesis that ANGPTL3 acts to reduce overall lipoprotein assembly and secretion in the liver will be tested directly by comparing the production rates of VLDL1, VLDL2, IDL and LDL apoB100, and the secretion rate of VLDL1-TG and VLDL2-TG in the three subject groups.

Further outcomes will be to align the proteomic and lipidomic compositional data with variation in kinetic parameters. If it is the case that ANGPTL3 LOF carriers have very low levels of remnant particles (and other atherogenic lipoproteins) then the composition of VLDL fractions, IDL and LDL may reveal a 'low risk signature' that is helpful when evaluating the efficacy of agents designed to lower or inhibit ANGPTL3 action.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited on the basis of their known status for the S17X LOF variant.
* Inhabitants of the Campodimele village, near Rome, Italy
* Homozygotes for ANGPTL3 S17X variant OR
* Heterozygotes having:
* ANGPTL3 plasma levels (<150ng/ml) AND
* TG (<120mg/dl).
* Healthy controls

Exclusion Criteria:

* NYHA > II or MACE in the previous 6 months
* CKD > stage III
* Uncontrolled hypertension BP > 160/100 mmHg
* Hypercholesterolemia (LDL> 190 mg/dL)
* Hypertrigliceridemia (TGs> 900 mg/dL)
* Any lipid-lowering medication
* Uncontrolled type 2 Diabetes mellitus (HbA1c > 7,5%)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Lipoprotein Kinetics | 36 months
  Measure of deuterated leucine enrichment in apoB in lipoprotein fractions after an oral fat in temporized blood draws
Kinetics of TG in VLDL1 and VLDL2. | 36 months
  Measure of deuterium enrichent in TGs in VLDL1 and VLD2 fractions in temporized blood draws over the 5 days subsequent an oral fat load
Lipoprotein Proteomics | 36 months
  Protein determination and quantification in different lipoprotein fraction to establish a specific proteomic profile for ANGPTL3 deficient subjects which might be associated with low cardiovascular risk

IPD SHARING:
Plan to Share IPD: No